CLINICAL TRIAL: NCT04485442
Title: Patient Reported Outcome Measures After Treatment of Skin Cancers on the Face - a Pilot Study
Brief Title: Patient Reported Outcome Measures After Treatment of Skin Cancers on the Face
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00301; ch20Schaefer2
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Skin Cancer
Keywords: melanoma; SCC in the face; infiltrative basal cell carcinoma on the face; Mohs Surgery
MeSH Terms: conditions — Skin Neoplasms; Melanoma | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection by questionnaires — psychological well-being in patients evaluated by Patient Reported Outcomes (PRO)
Other: data collection (photos of the patients' tumors) — photos of the patients' tumors will be taken at baseline and at follow-up after the surgery

SUMMARY:
This study is to evaluate the psychological well-being in patients diagnosed with skin cancer (melanoma and Squamous Cell Carcinoma (SCC) in the face) at the time of diagnosis and after treatment. Patients diagnosed with primary melanoma and/or SCC and/or infiltrative basal cell carcinoma on the face subjected to surgical treatment (excision or Mohs Surgery) will be included. All patients will receive questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with melanoma, SCC and/or infiltrative basal cell carcinoma on the face for surgical treatment and planned for excision or Mohs surgery
* patients who are able to give informed consent

Exclusion Criteria:

* Electrodesication and curettage of the tumour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with melanoma, SCC and /or infiltrative basal cell carcinoma on the face are eligible for the study and will be recruited at the Department of Dermatology and Plastic Surgery at University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in Belastungs-Thermometer questionnaire | at Screening Visit (V1), V3 (7 days post surgery), V4 (90 days post surgery), V5 (180 days post surgery), V6 (360 days post surgery)
  extent of distress on a scale from 0-10 (0=no distress, 10=extremely distress).

SECONDARY OUTCOMES:
Change in European Organization for Research and Treatment of Cancer (EORTC-QLQ-C30) questionnaire | at Screening Visit (V1), V3 (7 days post surgery), V4 (90 days post surgery), V5 (180 days post surgery), V6 (360 days post surgery)
  TheEORTC- QLQ-C30 is composed of both multiitem scales and single-item measures. These include 5 functional scales (cognitive, CF; emotional, EF; physical, PF; role, RF; and social functioning, SF), 3 symptom scales (fatigue, FA; nausea/vomiting, NV; and pain, PA), a global health status/QoL scale and 5 single items assessing additional symptoms (appetite loss, AP; constipation, CO; diarrhea, DI; dyspnea, DY; and sleep disturbance, SL) and perceived financial impact, FI. Each of the multiitem scales includes a different set of items-no item occurs in more than 1 scale. All of the scales and single-item measures range in score from 0-100. A high scale score represents a higher response level.
Change in WHO-DAS questionnaire | at Screening Visit (V1), V3 (7 days post surgery), V4 (90 days post surgery), V5 (180 days post surgery), V6 (360 days post surgery)
  The WHO-DAS measures items in six domains of functioning as experienced over the past 30 days: mobility, self-care, life activities, understanding and communicating (U&C), interpersonal interactions, and participation in society. The 12-item tool assesses each domain with two items that are measured on a 3-point scale in which 1 indicates no disability, 2 indicates mild to moderate disability, and 3 indicates severe to extreme disability. These items were summed to generate a total score between 12 (no disability) and 36 (maximum disability).
Change in FACE-Q questionnaire | at Screening Visit (V1), V3 (7 days post surgery), V4 (90 days post surgery), V5 (180 days post surgery), V6 (360 days post surgery)
  The FACE-Q questionnaire measures three overarching domains: facial appearance, quality of life and experience of care over the past 7 days. The FACE-Q Skin Cancer Module is composed of 56 items with scales from 1-4 which range in scoring from 0-100. The FACE-Q Skin Cancer module includes two quality of life scales measuring appearance-related distress and skin cancer worry. Additionally, the participants will be asked about skin protection behaviours and adverse events following the skin cancer treatment. The FACE-Q appearance scale consists of satisfaction with the appearance of the face overall and how bothered a patient is by facial scars
Change in photos of the patients' tumors | at Screening Visit (V1), V3 (7 days post surgery), V4 (90 days post surgery), V5 (180 days post surgery), V6 (360 days post surgery)
  Change in photos of the patients' tumors

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J Schaefer, Prof. Dr. med., Principal Investigator — Department of Plastic, Reconstructive and Aesthetic Surgery, University Hospital Basel
Locations (1):
- Department of Plastic, Reconstructive and Aesthetic Surgery and Department of Dermatology , University Hospital Basel, Basel, Switzerland